CLINICAL TRIAL: NCT02878551
Title: Evaluation of the Benefits of a Program of Prehabilitation: Pilot Study
Brief Title: Evaluation of the Benefits of a Prehabilitation Program : Pilot Study
Acronym: PrehabPilote
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hopital Foch (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016/29; 2016-A00981-50 (Other: ANSM)
Record Dates: First submitted 2016-08-22; First posted 2016-08-25 (Estimated); Last update posted 2021-03-09 (Actual); Status verified 2021-03

CONDITIONS: Surgery; Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prehabilitation program (Experimental): Multimodal prehabilitation intervention composed of exercise, nutritional supplement and psychological well-being
  Interventions: Other: Prehabilitation program

INTERVENTIONS:
Other: Prehabilitation program — multimodal prehabilitation intervention composed of exercise, nutritional supplement and psychological well-being

SUMMARY:
The process of enhancing functional capacity of the individual in anticipation of an upcoming stressor has been termed "prehabilitation". In the present pilot trial, the impact of a multimodal prehabilitation intervention composed of exercise, nutritional supplement and psychological well-being begun in the preoperative period will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old
* Affiliated with a social security system
* Having indicated their non-opposition
* Must undergo a surgical intervention within a period of at least one month after the completion of the initial inclusion assessment and / or chemotherapy and / or radiotherapy

Non-inclusion criteria:

* Refusal of participation
* Pregnant or breastfeeding woman
* Inability to walk or initial physical assessment
* Patient under guardianship or curatorship
* Inability to complete questionnaires

Exclusion criteria:

* Cognitive disorders detected by the geriatric consultation
* Lost
* Death before surgery or chemotherapy or radiotherapy
* Shortened preoperative preparation time (<18 days)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-10-07 (Actual); Primary Completion 2017-06-23 (Actual); Study Completion 2017-06-23 (Actual)

PRIMARY OUTCOMES:
6 minutes walk test | 7 months

CONTACTS AND LOCATIONS:
Overall Officials: Morgan Le Guen, MD, Principal Investigator — Hopital Foch
Locations (1):
- Hopital Foch, Suresnes, France

IPD SHARING:
Plan to Share IPD: No